CLINICAL TRIAL: NCT01284608
Title: Metabolic Changes in Prostate Cancer Patients With Androgen-ablation Therapy (AAT)
Acronym: UROCOR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OES-DUM-2010/1
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Prostatic Cancer
Keywords: Observational; prospective; metabolic changes; metabolic syndrome; diabetes; prostatic cancer; risk fracture
MeSH Terms: conditions — Prostatic Neoplasms; Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational, prospective, non-interventional and multi-centre study, to assess the impact of androgen ablation therapy in blood triglycerides, cholesterol and glucose, body fat distribution and fracture risk to ten years using FRAX model in patients with prostate cancer. The patients will be following for 12 months

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patient requiring androgen-ablation treatment: LHRH analogs, surgical castration, antiandrogen treatment
* Provision of informed consent prior to conducting any study-related procedure

Exclusion Criteria:

* Patient involved in a Clinical Trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients in androgen-ablaction treatment in urological departments
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome | 3 months
Metabolic syndrome | 6 months
Metabolic syndrome | 12 months
Diabetes | 3 months
Diabetes | 6 months
Diabetes | 12 months

SECONDARY OUTCOMES:
Fracture Risk Assessment Tool (FRAx) assessment | 0 and 12 months

CONTACTS AND LOCATIONS:
Locations (33):
- Spain (33):
  - Research Site, Albacete, Albacete
  - Research Site, El Ejido, Almeria
  - Research Site, Huercal Overa, Almeria
  - Research Site, Mérida, Badajoz
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Barcelona, Barcelona
  - Research Site, El Hospitalet de Llobregat, Barcelona
  - Research Site, Sabadell, Barcelona
  - Research Site, Aranda de Duero, Burgos
  - Research Site, Miranda de Ebro, Burgos
  - Research Site, Córdoba, Cordoba
  - Research Site, Ferrol, Coru?a
  - Research Site, Granada, Granada
  - Research Site, Guadalajara, Guadalajara
  - Research Site, Donostia / San Sebastian, Guipuzcoa
  - Research Site, Jaén, Jaen
  - Research Site, Logroño, La Rioja
  - Research Site, Monforte (casco Urbano), Lugo
  - Research Site, Alcalá de Henares, Madrid
  - Research Site, Coslada, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Majadahonda, Madrid
  - Research Site, San Sebastián de los Reyes, Madrid
  - Research Site, Antequera, Malaga
  - Research Site, Vigo, Pontevedra
  - Research Site, Osuna, Sevilla
  - Research Site, Reus, Tarragona
  - Research Site, Toledo, Toledo
  - Research Site, Barakaldo, Vizcaya
  - Research Site, Bilbao, Vizcaya
  - Research Site, Galdakao, Vizcaya
  - Research Site, Calatayud, Zaragoza
  - Research Site, Zaragoza, Zaragoza